CLINICAL TRIAL: NCT03190655
Title: Efficacy and Safety of Aluminaid Versus Hydrogel Wound Dressings in the Treatment of Partial Thickness Burns
Brief Title: Efficacy and Safety of Aluminaid Versus Hydrogel Wound Dressings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped by the Sponsor due to their change in product development priorities.
Sponsor: Melva Louisa (Other)
Responsible Party: Sponsor-Investigator, Melva Louisa, Trial Director, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aluminaid
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Partial-thickness Burn
MeSH Terms: interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: Patients who attend the clinical sites, presenting with untreated partial thickness burns less than 4 hours, and meet the inclusion and exclusion criteria
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The person that assess the degree of epithelization will be presented with photos of the burn conditions and will not be given information of the patient's treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aluminaid (Experimental): Treatment group: Aluminaid wound dressing
  Interventions: Device: Aluminaid
- Hydrogel (Active Comparator): Hydrogel wound dressing (Trademark: Burnshield)
  Interventions: Device: Hydrogel

INTERVENTIONS:
Device: Aluminaid — Aluminaid wound dressings is a hydrogel based wound dressing that is integrated with aluminium
  Arms: Aluminaid
Device: Hydrogel — Hydrogel based wound dressing
  Arms: Hydrogel

SUMMARY:
Burn injury is the result of an energy transfer that destroys the skin and adjacent tissues. Partial thickness burn wounds are painful and difficult to manage. The aim of burn treatment in partial thickness burns is to promote rapid wound healing, decrease pain, protect wound from infections, minimize scar formation and functional impairment In recent years, there are progressive development of new dressing material with a variety of option for depth adapted wound management. Many wound dressings are available for superficial and partial thickness burns. Hydrogel based wound dressing provides good biocompatibility with the skin and mucosa and promotes hydration of the wound bed.

Aluminaid wound dressings is a hydrogel based wound dressing that is integrated with aluminium that was designed to reduce acute pain in the treatment of superficial and partical thickness burn injuries.

Up to date, no evidence regarding integrated with aluminium sheet in hydrogel based wound dressings for the use in partial thickness burns. Therefore this trials is aimed to evaluate the efficacy and safety of Aluminaid versus Hydrogel for the treatment of partial thickness burns.

DETAILED DESCRIPTION:
This is a prospective, randomized, open label, active controlled trial that aim to evaluate the efficacy and safety of Aluminaid versus Hydrogel wound dressings in the treatment of partial thickness burns.

The study is a multi center trial in children and adults of 12 - 65 years old with partial thickness burns.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children of 12 - 65 years old
* Partial thickness thermal burns of minimally 1% total body surface area (TBSA)
* Admission of less than 4 hours of burn injury
* Patients/legal guardian still have the ability to undergo examinations and give written informed consent.

Exclusion Criteria:

* Total body surface area (TBSA) of more than 20%
* Burns caused by chemicals, electricity or radiation
* Superficial and partial thickness burns located on the faces, palms, soles, genitalia, perineum and joint areas
* Superficial and partial thickness burns with compartment syndrome
* Superficial and partial thickness burns with a history of life-threatening trauma
* Had concomitant disease such as diabetes mellitus
* Signs of infected burns
* Patients with known allergies to product containing aluminium, hydrogel or a history of contact dermatitis
* Other conditions which according to the investigator's judgment are not appropriate to be included in the study.
* Treated with other agents before attend to clinic (oil, tooth paste, betadine, rivanol etc)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Wound healing | Up to 21 days
  Wound healing as determine by the time of complete re-epithelization of the study area, in days.

SECONDARY OUTCOMES:
Erythema | at the time of admission up to 30 minutes
  The presence of erythema
Bullae | at the time of admission up to 30 minutes
  The presence of bullae
Pain score | At the time of admission up to 30 minutes and 1st week of follow up
  Pain score is determined by VAS score (1 - 10: 1 is no pain 10 is severe pain).
Adverse events | At the time of admission up to 21 days of follow up
  The adverse events in patients treated with Aluminaid versus Hydrogel as determined by the proportion of patients who experience adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wawaimuli Arozal, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Clinic of Clinical Research Supporting Unit, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grippaudo FR, Carini L, Baldini R. Procutase versus 1% silver sulphadiazine in the treatment of minor burns. Burns. 2010 Sep;36(6):871-5. doi: 10.1016/j.burns.2009.10.021. Epub 2010 Jan 15. PMID 20079572
- [Background] Cancio LC, Lundy JB, Sheridan RL. Evolving changes in the management of burns and environmental injuries. Surg Clin North Am. 2012 Aug;92(4):959-86, ix. doi: 10.1016/j.suc.2012.06.002. PMID 22850157
- [Background] Hettiaratchy S, Dziewulski P. ABC of burns: pathophysiology and types of burns. BMJ. 2004 Jun 12;328(7453):1427-9. doi: 10.1136/bmj.328.7453.1427. No abstract available. PMID 15191982
- [Background] Lars PK, Giretzlehner M, Trop M, Parvizi D, Spendel S, Schintler M, Justich I, Wiedner M, Laback C, Lumenta DB. The properties of the "ideal" donor site dressing: results of a worldwide online survey. Ann Burns Fire Disasters. 2013 Sep 30;26(3):136-41. PMID 24563639
- [Background] Rowan MP, Cancio LC, Elster EA, Burmeister DM, Rose LF, Natesan S, Chan RK, Christy RJ, Chung KK. Burn wound healing and treatment: review and advancements. Crit Care. 2015 Jun 12;19:243. doi: 10.1186/s13054-015-0961-2. PMID 26067660
- [Background] Selig HF, Lumenta DB, Giretzlehner M, Jeschke MG, Upton D, Kamolz LP. The properties of an "ideal" burn wound dressing--what do we need in daily clinical practice? Results of a worldwide online survey among burn care specialists. Burns. 2012 Nov;38(7):960-6. doi: 10.1016/j.burns.2012.04.007. Epub 2012 May 8. PMID 22571855
- [Background] Serrano C, Boloix-Tortosa R, Gomez-Cia T, Acha B. Features identification for automatic burn classification. Burns. 2015 Dec;41(8):1883-1890. doi: 10.1016/j.burns.2015.05.011. Epub 2015 Jul 15. PMID 26188898
- [Background] Wasiak J, Cleland H, Campbell F, Spinks A. Dressings for superficial and partial thickness burns. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD002106. doi: 10.1002/14651858.CD002106.pub4. PMID 23543513